CLINICAL TRIAL: NCT05747716
Title: SBRT Combined With Fruquintinib Plus PD-1/CTLA-4 Antibody Cadonilimab for Third-line Treatment in Metastatic Colonrectal Cancer.
Brief Title: SBRT Combined With Fruquintinib Plus PD-1/CTLA-4 Antibody for Third-line Treatment in mCRC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCRC-3
Record Dates: First submitted 2023-02-18; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT, Fruquintinib, Cadonilimab (Experimental)
  Interventions: Drug: SBRT, Fruquintinib, Cadonilimab

INTERVENTIONS:
Drug: SBRT, Fruquintinib, Cadonilimab — Radiation: Stereotactic body radiationtherapy (SBRT) for metastatic sites (less than 5) Fruquintinib: 5mg, po, everyday; Cadonilimab: 10mg/kg, iv, q3w

SUMMARY:
The study is a phase II clinical study. The purpose of the study is to evaluate the efficacy and safety of SBRT combined with Fruquintinib Plus PD-1/CTLA-4 Antibody for Third-line Treatment in mCRC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy proven unresectable MCRC.
2. Patients must have received first-line and second-line chemotherapy, and approved a progressive disease.
3. Age ≥ 18 years
4. Patients must have measurable disease at baseline.
5. Patients can have up to only 5 discrete active extracranial lesions (≤3 in the liver and ≤3 in the lung) identified by position-emission tomography (PET) scan and also seen on correlative plain film, CT scan, or MRI within 8 weeks prior to the initiation of radiotherapy.
6. Patients who previously received radiotherapy to the primary site will be ineligible if there is CT evidence of disease progression within the past 3 months.
7. Patients must have a Karnofsky Performance Scores (KPS) >60 8. Aspartate aminotransferase, alanine aminotransferase & Alkaline phosphates must be ≤ 2.5 times the upper limit of normal (ULN). Total bilirubin must be within the limit of normal.

9. Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm3. 10. Patients should have adequate renal function (serum creatinine ≤1.5 times the ULN). 11. Females of childbearing potential should have a negative pregnancy test. 12. Patients who would be receiving radiation for lung lesions who are known or suspected by the treating radiation oncologist to have compromised lung function must have a documented forced expiratory volume in 1 second (FEV1) ≥ 1 litre.

13. Patients must provide verbal and written informed consent to participate in the study.

14. Total bilirubin: within normal institutional limits

Exclusion Criteria:

1. Patients with either untreated brain metastases or brain metastases treated within the past three months are ineligible
2. Patients with serious, uncontrolled, concurrent infection(s).
3. Significant weight loss (>10%) in the prior 3 months.
4. Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cancers.
5. Patients with more than 5 discrete metastatic lesions.
6. Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
7. Unwillingness to participate or inability to comply with the protocol for the duration of the study.
8. Patients who are pregnant. Patients with reproductive capability will need to use adequate contraception during the time of participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Progression free survival

SECONDARY OUTCOMES:
Actuarial rate in-field local control | 2 years
  To describe the actuarial rate in-field local control and rate of out-of-field disease progression
Toxicities | 2 years
  Acute toxicity was scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0 criteria during and up to 3 months after radiotherapy. Late toxicity was graded using the Radiation Therapy Oncology Group (RTOG)/European Organisation for the Research and Treatment of Cancer (EORTC) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China